CLINICAL TRIAL: NCT01056003
Title: Gastric Inlet Patches of the Cervical Esophagus. Incidental Finding or Underrated Cause of Globus Sensations.
Brief Title: Prevalence of Gastric Inlet Patches of the Cervical Esophagus.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Collaborators: Institut für Allgemeine Pathologie und Pathologische Anatomie der TU München (Unknown); Klinik für Kinder und Jugendmedizin, Klinikum Dritter Orden; München (Unknown); Klinik für Kinder und Jugendmedizin, Universitätsklinikum Ulm (Unknown); Kinderklinik im Dr. von Haunerschen Kinderspital, Universität München (Unknown)
Responsible Party: Monther Bajbouj, MD, Klinikum rechts der Isar, Technische Universitaet Munich
Other Study IDs: Gips in Kids
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Association of Heterotopic Gastric Mucosa of the Cervical Esophagus and Globus Sensations
Keywords: gastric inlet patch; prevalence; globus sensations
MeSH Terms: conditions — Globus Sensation | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- all patients admitting endoscopy for EGD
  Interventions: Other: Endoscopy

INTERVENTIONS:
Other: Endoscopy — observational endoscopy in all patients an EGD is planned anyway

SUMMARY:
As known from several observational and retrospective endoscopic studies the prevalence of gastric inlet patches (GIPs) of the cervical esophagus is estimated between 1-10%. In most cases GIPs are found within endoscopy as an incident finding, since in most cases they are harmless and do not cause any symptoms. None the less several data exist where an association between GIPs and globus sensations is discussed. Case reports even refer to bleeding complications and moreover to malignant transformations of GIPs.

As a result of the assumed association of GIPs and globus sensations we performed a pilot trial. Here we included 10 patients with globus and GIPs and were able to demonstrate a significant symptom relief after ablation of the GIP (Meining et al, Endoscopy 2006). To exclude a potential placebo-effect we concluded a multicenter and sham controlled trial where we imposingly were able to prove the symptom relief after ablation of the GIPs (Bajbouj et al, Gastroenterology 2009).

All patients, who are scheduled for esophagogastroduodenoscopy (EGD) in any of the above mentioned endoscopical departments are routinely standardized asked whether they have any hints suggestive for globus sensations (modified globus-questionnaire from Deary et al., J Psychosom Res 1995). Concurrently it is noted, whether the patients have endoscopical detected GIP. All GIPs are biopsied and examined in one institute. Together with anamnestic data (age, gender) a talley sheet gives a survey of all relevant information to prove or disprove following hypotheses.

Study hypotheses:

1. The presence of GIPs is associated with globus sensations. In other words: Do patients with globus sensations significantly more often have GIPs?
2. GIPs are not congenital, they arise in the course of the time and become symptomatic. In other words: Do GIPs significantly occur in more elderly people?
3. The more increased the GIPs diameter is the more likely globus sensations are present? In other words: Do huge GIPs cause significantly more often symptoms than small ones?
4. The more mucus-producing mucosa is histologically proven the more likely globus sensations are present? In other words: Do we find more cardiac mucosa in patients with symptoms than fundus mucosa?

ELIGIBILITY:
Exclusion Criteria:

* emergency EGD
* any condition which contraindicates biopsy sampling
* unavailable informed consent for the GD

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients admitting one of the above mentioned endoscopic departments for a scheduled EGD
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Monther Bajbouj, MD, Principal Investigator — Technical University Munich; Sybille Koletzko, Professor, Principal Investigator — Kinderklinik im Dr. von Haunerschen Kinderspital, Universität München; Slim Saadi, MD, Principal Investigator — Klinik für Kinder und Jugendmedizin, Klinikum Dritter Orden; München; Susanne Liptay, MD, Principal Investigator — Technical University Munich; Carsten Posovsky, Principal Investigator — University Ulm
Locations (1):
- Klinikum rechts der Isar, Munich, Bavaria, Germany

REFERENCES:
- [Result] Bajbouj M, Becker V, Eckel F, Miehlke S, Pech O, Prinz C, Schmid RM, Meining A. Argon plasma coagulation of cervical heterotopic gastric mucosa as an alternative treatment for globus sensations. Gastroenterology. 2009 Aug;137(2):440-4. doi: 10.1053/j.gastro.2009.04.053. Epub 2009 May 4. PMID 19410576
- [Result] Meining A, Bajbouj M, Preeg M, Reichenberger J, Kassem AM, Huber W, Brockmeyer SJ, Hannig C, Hofler H, Prinz C, Schmid RM. Argon plasma ablation of gastric inlet patches in the cervical esophagus may alleviate globus sensation: a pilot trial. Endoscopy. 2006 Jun;38(6):566-70. doi: 10.1055/s-2006-925362. PMID 16802267